CLINICAL TRIAL: NCT02331992
Title: Positive Airway Pressure Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CIA-146
Record Dates: First submitted 2015-01-04; First posted 2015-01-06 (Estimated); Results first posted 2018-10-29 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Continuous Positive Airway Pressure
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive airway pressure adherence program (Experimental): Participants will be enrolled in the automated adherence program and will receive supportive messages while they use CPAP as prescribed by their healthcare provider. These messages are designed to aid the participant towards therapy adherence.
  Interventions: Behavioral: Adherence program

INTERVENTIONS:
Behavioral: Adherence program — Participants will receive supportive messages while enrolled in the program.

SUMMARY:
Obstructive Sleep Apnea (OSA) is a common sleep disordered breathing condition effecting around 2-4% of the middle aged population and is characterized by periodic collapse of the upper airway during sleep. Continuous Positive Airway Pressure (CPAP) is the primary treatment for patients with OSA. Despite the effectiveness of CPAP in abolishing upper airway obstruction, acceptance of and adherence with therapy has been sub-optimal.

Over the past decade, considerable research has focused on determining the factors responsible for poor CPAP adherence. Two key areas have been identified: patient-reported symptoms, including mask discomfort, pressure intolerance and nasal symptoms and the importance of patient education and support. In addition we know that the patient experience during the crucial first days and weeks of their journey predicts longer term adherence.

This study investigates the ability of an automated program that assists patients towards continuous positive airway pressure (CPAP) therapy adherence.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18years of age
* Diagnosed with OSA (AHI >5 events/hour) and eligible for CPAP (fixed or auto) treatment under local requirements
* Naïve to CPAP therapy, i.e. have not been prescribed CPAP in the past 5 years
* Own a mobile phone, and has reliable mobile network coverage at their home.
* Either: the participant will use a modem; OR the participant has access to a home internet connection (either their own, or a neighbours or friend etc) and is willing to perform a home upload.

Exclusion Criteria:

* Contraindicated for CPAP therapy
* Medically unstable condition/diagnosis that is not yet under control
* Co-existing sleep disorder (however clinically diagnosed insomnia can be included in the study)
* Periodic Limb Movement Arousal Index (PLMA) greater than 15/hr during the diagnostic study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-02; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamish Collie, MHlthSc, Study Chair — Fisher & Paykel Healthcare
Locations (3):
- United States (3):
  - Alabama Sleep Clinic, Huntsville, Alabama
  - IV Care & Respiratory, Belleville, Illinois
  - SleepMed of South Carolina, Columbia, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Airway Pressure Adherence Program
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Positive Airway Pressure Adherence Program
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 44 [26 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Participant Providing Feedback
Description: Participants will be provided questionnaires so as to provide program feedback.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Airway Pressure Adherence Program
Number analyzed (Participants) | 34
Participants | 26

2. Secondary Outcome: Healthcare Provider Feedback
Description: Healthcare providers will be provided questionaires so as to provide program feedback.
Time Frame: 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Positive Airway Pressure Adherence Program
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Positive Airway Pressure Adherence Program
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 1/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Positive Airway Pressure Adherence Program (N=34)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agrees to supply the sponsor with any proposed publications or presentation. Any information that affect the sponsor IP, or information that is commercially sensitive, may be delayed, deleted or amended.